CLINICAL TRIAL: NCT01838616
Title: Evaluation of the Effectiveness, Safety, and Tolerability of Tapentadol PR Versus Oxycodone/Naloxone PR in Non-opioid Pre-treated Subjects With Uncontrolled Severe Chronic Low Back Pain With a Neuropathic Pain Component.
Brief Title: Tapentadol Prolonged Release (PR) Versus Oxycodone/Naloxone Prolonged Release in Severe Chronic Low Back Pain With a Neuropathic Component.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF5503/60; 2012-002943-11 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Back Pain; Low Back Pain; Neuropathic Pain
Keywords: Severe chronic low back pain; Neuropathic pain; Constipation
MeSH Terms: conditions — Back Pain; Low Back Pain; Neuralgia; Constipation | interventions — Tapentadol; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol Prolonged Release (PR) (Experimental)
  Interventions: Drug: Tapentadol Prolonged Release
- Oxycodone/Naloxone Prolonged Release (Active Comparator)
  Interventions: Drug: Oxycodone/Naloxone Prolonged Release

INTERVENTIONS:
Drug: Tapentadol Prolonged Release — All participants started with 50 mg tapentadol hydrochloride prolonged release (twice daily). The dose of tapentadol hydrochloride prolonged release will be adjusted in increments of 50 mg to a level that provided adequate analgesia. Titration will be after a minimum of 3 days on a dose. Participants are permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). After titration participants will remain on the stable dose for 9 weeks.
  Other Names: Nucynta; Palexia
  Arms: Tapentadol Prolonged Release (PR)
Drug: Oxycodone/Naloxone Prolonged Release — All participants start with 10 mg/5 mg oxycodone/naloxone (twice daily). The dose of oxycodone/naloxone may be adjusted in increments of 10mg/ 5 mg oxycodone/naloxone to a level that provide adequate analgesia. Titration will be after a minimum of 3 days on a dose. Participants will be permitted a maximum dose of 50 mg/ 20 mg oxycodone/naloxone twice daily a day (100 mg/40 mg total daily dose). After titration participants will remain on the stable dose for 9 weeks.
  Other Names: Targin
  Arms: Oxycodone/Naloxone Prolonged Release

SUMMARY:
This was a clinical effectiveness trial designed to compare the effectiveness, safety, and tolerability of treatment with tapentadol prolonged release with that of oxycodone/naloxone prolonged release in non-opioid pre-treated subjects with severe chronic low back pain with a neuropathic pain component.

Both tapentadol and the opioid oxycodone are effective in chronic severe pain and tapentadol and oxycodone/naloxone have shown advantages in gastrointestinal tolerability versus oxycodone. Therefore, it was of high scientific interest to compare the latter 2 analgesics with respect to gastrointestinal tolerability. Tapentadol may have advantages regarding the neuropathic pain-related symptoms of low back pain due to its 2 mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Male or female 18 years of age or older.
* Women of childbearing potential must have a negative pregnancy test at the Enrollment Visit.
* Women of childbearing potential must practice medically acceptable methods of birth control during the trial.
* Participant must be appropriately communicative and able to differentiate with regard to location and intensity of the pain, and to complete the questionnaires used in this trial.
* Participants must have a diagnosis of chronic low back pain; chronic pain defined as pain lasting for at least 3 months prior to enrollment.
* Participant's pain must require a strong analgesic (defined as World Health Organization Step III) as judged by the investigator.
* Participants who require a washout of co-analgesics at enrolment must have an average pain score (NRS-3) of 5 points or higher. Participants who do not require a washout of co-analgesics at enrollment must have an average pain intensity score (NRS-3) during the last 3 days of 6 points or higher.
* The painDETECT diagnostic screening questionnaire must be either "positive" (score of 19 to 38 inclusive) or "unclear" (score of 13 to 18 inclusive). If the participant is being treated with a stable regimen of centrally acting co-analgesics, a "negative" painDETECT score (score 9 points or higher).

Inclusion criteria prior to allocation to treatment:

* Participants must have an average pain intensity score (NRS-3) during the last 3 days of 6 points or higher.
* Participants must score either "positive" (score of 19 to 38 inclusive) or "unclear" (score of 13 to 18 inclusive) on the painDETECT diagnostic screening questionnaire.

Exclusion Criteria:

* Presence of a clinically significant disease or clinical laboratory values that in the investigator's opinion may affect effectiveness, quality of life, or safety/tolerability assessments.
* Presence of active systemic or local infections that may, in the opinion of the investigator, affect the effectiveness, quality of life, or safety/tolerability assessments.
* Employees of the investigator or trial site, with direct involvement in this trial or other trials under the direction of the investigator or trial site, as well as family members of employees of the investigator.
* Participation in another trial concurrently, or within 4 weeks prior to the Enrollment Visit.
* Known to or suspected of not being able to comply with the protocol and/or appropriate use of the Investigational Medicinal Products.
* Any painful procedures (e.g., major surgery) scheduled during the trial duration (Enrollment Visit until Final Evaluation Visit) that may, in the opinion of the investigator, affect the effectiveness, quality of life, or safety assessments.
* Pending litigation or application for insurance/governmental benefits due to chronic pain or disability and/or if the granted benefits might be influenced by a successful participation in the trial.
* Low back pain caused by cancer and/or metastatic diseases.
* History of alcohol or drug abuse, or suspicion thereof in the investigator's judgment.
* Presence of concomitant autoimmune inflammatory conditions.
* Participants with acute intoxication with alcohol, hypnotics, centrally acting analgesics, or psychotropic active substances.
* Participants with severe renal impairment, i.e., estimated glomerular filtration rate less than 30 mL/min (according to the National Kidney Foundation 2002).
* Known history of clinical laboratory values or current clinical laboratory values reflecting moderately or severely impaired hepatic function.
* History of seizure disorder or epilepsy.
* Any of the following within 1 year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm (including brain metastases if present at the Enrollment Visit). Severe traumatic brain injury within 15 years (consisting of 1 or more of the following: brain contusion, intracranial hematoma, either unconsciousness or post traumatic amnesia lasting more than 24 hours) or residual sequelae suggesting transient changes in consciousness.
* Pregnant or breast-feeding women.
* Severe respiratory depression with hypoxia and/or hypercapnia, acute or severe bronchial asthma or severe chronic obstructive pulmonary disease.
* Presence or suspicion of paralytic ileus.
* Participants with severe cardiac impairment, e.g., New York Heart Association class >3, myocardial infarction less than 6 months prior to the Enrollment Visit, and/or unstable angina pectoris and/or cor pulmonale.
* Participant with known history of rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.
* History of allergy or hypersensitivity to tapentadol, oxycodone, naloxone, and their formulations.
* Participants with acute biliary obstruction or acute pancreatitis.
* Participants with hypothyroidism (including myxedema) or Addison's disease.
* Participants taking any prohibited concomitant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (50):
- Austria (2):
  - AT001, Senftenberg
  - AT002, Vienna
- Germany (33):
  - DE005, Bad Saarow
  - DE007, Berlin
  - DE021, Berlin
  - DE009, Berlin
  - DE030, Berlin
  - DE020, Bochum
  - DE023, Böhlen
  - DE029, Cologne
  - DE008, Cologne
  - DE028, Cottbus
  - DE012, Dresden
  - DE032, Essen
  - DE017, Frankfurt
  - DE003, Frankfurt
  - DE011, Görlitz
  - DE031, Hamburg
  - DE013, Hanover
  - DE001, Kiel
  - DE027, Kiel
  - DE014, Kiel
  - DE004, Leipzig
  - DE034, Leipzig
  - DE018, Leipzig
  - DE015, Magdeburg
  - DE006, Mainz
  - DE002, Mittweida
  - DE010, Rudolstadt
  - DE025, Schwerin
  - DE019, Stadtroda
  - DE016, Weinheim
  - DE024, Westerstede
  - DE026, Wiesbaden
  - DE022, Wiesbaden
- Italy (5):
  - IT003, Catania
  - IT001, Genova
  - IT002, Parma
  - IT004, Pavia
  - IT005, Varese
- Spain (10):
  - ES006, A Coruña
  - ES007, Barcelona
  - ES001, Barcelona
  - ES003, Centelles
  - ES008, Guadix
  - ES002, Madrid
  - ES010, Madrid
  - ES009, Madrid
  - ES004, Oviedo
  - ES005, Santiago de Compostela

REFERENCES:
- [Result] Baron R, Likar R, Martin-Mola E, Blanco FJ, Kennes L, Muller M, Falke D, Steigerwald I. Effectiveness of Tapentadol Prolonged Release (PR) Compared with Oxycodone/Naloxone PR for the Management of Severe Chronic Low Back Pain with a Neuropathic Component: A Randomized, Controlled, Open-Label, Phase 3b/4 Study. Pain Pract. 2016 Jun;16(5):580-99. doi: 10.1111/papr.12308. Epub 2015 Jun 12. PMID 26095455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 22 Mar 2013 with the enrollment of the first participant and was completed on 28 Jan 2014 when the last subject completed the last follow-up examination according to the protocol.
Pre-assignment Details: 367 participants signed informed consent. 89 participants did not meet the inclusion/exclusion criteria, 16 participants withdrew and 4 participants left the trial for other reasons.
  Participants randomized to oxycodone/naloxone PR could be switched to tapentadol PR treatment in the pick-up arm of the trial.
Groups:
- Tapentadol Prolonged Release: All participants started with 50 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted in increments of 50 mg to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
- Oxycodone/Naloxone Prolonged Release: All participants started with 10 mg/5 mg oxycodone/naloxone prolonged release (twice daily). The dose of oxycodone/naloxone prolonged release could be adjusted in increments of 10 mg/5 mg oxycodone/naloxone to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 50 mg/20 mg oxycodone/naloxone twice daily (100 mg/40 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
Period: Titration Period
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Started | 130 | 128
No Post Baseline Pain Intensity Values | 0 | 2
Major Protocol Deviations | 13 | 16
Switched to Pick-up Arm | 0 | 43
Full Analysis Set | 130 | 128
Per Protocol Set | 117 | 112
Completed | 100 | 62
Not Completed | 30 | 66
Not completed — Adverse Event | 18 | 48
Not completed — Lack of Efficacy | 5 | 12
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Technical problems | 1 | 0
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 0 | 1
Period: Continuation Period
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Started | 100 | 62
Switched to Pick-up Arm | 0 | 7
Completed | 86 | 48
Not Completed | 14 | 14
Not completed — Lack of Efficacy | 3 | 5
Not completed — Adverse Event | 8 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Technical problems | 0 | 1
Period: Pick-up Arm
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Started | 50 (Switch to Tapentadol (PR) after Oxycodone/Naloxone (PR) treatment discontinuation.) | 0
Full Analysis Set | 49 | 0
Completed | 35 (Participants completed the tapentadol pick-up arm after initially on oxycodone/naloxone PR treatment) | 0
Not Completed | 15 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Technical problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release | Total
Number analyzed (Participants) | 130 | 128 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.48) | 58.4 (12.23) | 58.2 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 84 | 161
  Male | 53 | 44 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 130 | 128 | 258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 20 | 19 | 39
  Austria | 8 | 9 | 17
  Germany | 102 | 100 | 202
Dermatol pain present [Number; unit: participants] | 121 | 111 | 232
Lumbar radiculopathy [Number; unit: participants] | 76 | 75 | 151
Duration of pain [months] [Median (Full Range); unit: months] | 61.5 [4 to 552] | 72 [3 to 504] | 70.5 [3 to 552]
Height [Mean (Standard Deviation); unit: centimeters] | 168.9 (11.00) | 167.7 (9.71) | 168.3 (10.38)
Weight [Mean (Standard Deviation); unit: kilogram] | 85.3 (18.23) | 81.6 (18.43) | 83.5 (18.39)
painDETECT [Number; unit: participants] — The painDETECT questionnaire was used to determine the possibility of the presence of a neuropathic pain component. It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear". Participants being treated with a stable regimen of centrally acting co-analgesics at baseline were permitted if the score was at least 9.
  participants
    painDETECT positive | 96 | 97 | 193
    painDETECT unclear | 33 | 27 | 60
    painDETECT negative | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average Pain Intensity Score on an 11-point Numeric Rating Scale (NRS-3)
Description: For this pain assessment, the participant indicated the level of average pain experienced over the previous 3 days on an 11-point Numeric Rating Scale (NRS-3) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value reported represents the change from the randomization visit (i.e., the last 3 days in the washout period prior to Investigational Medicinal Product initiation and titration) to the end of the continuation period (i.e., up to 9 weeks on the stable dose). The theoretical values range from -10 to 10. A negative sign indicates a decrease in pain from the start of treatment. The higher the absolute values, the greater the change since the start of treatment (Baseline Visit).
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: The primary analysis was performed for the Per Protocol Set (PPS). Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Oxycodone/Naloxone Prolonged Release: All participants started with 10 mg/5 mg oxycodone/naloxone prolonged release (twice daily). The dose of oxycodone/naloxone prolonged release could be adjusted in increments of 10 mg/5 mg oxycodone/naloxone to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 50 mg/20 mg oxycodone/naloxone twice daily a day (100 mg/40 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 117 | 112
units on a scale | -3.7 (0.25) | -2.7 (0.26)

2. Primary Outcome: Change in the Patient Assessment of Constipation Symptoms (PAC-SYM) Total Score
Description: The Constipation Assessment (PAC-SYM) is a 12-item self-report questionnaire that assessed the severity of symptoms of constipation. Participants were asked "How severe have each of these symptoms been in the last two weeks?" e.g. "Pain in your stomach". There are 3 subscales: 4 questions on abdominal symptoms, 3 on rectal symptoms and 5 on stool symptoms. Responses were rated on a 5-point Likert scale ranging from 0 (absence of symptom) to 4 (very severe symptoms). If the changes in the overall or subscale scores are positive then there is a worsening in symptoms associated with constipation. The change in the assessment of constipation symptoms (PAC-SYM) total score from the Randomization Visit to the Final Evaluation Visit. The PAC-SYM overall score is the sum of scores of all non-missing items divided by the number of non-missing items (if at least 6 items were non-missing).
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: The primary analysis was performed for the Per Protocol Set (PPS).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 117 | 112
units on a scale | 0.07 (0.060) | 0.14 (0.062)

3. Secondary Outcome: Recalled Average Pain Intensity
Description: The recalled average pain intensity score on the NRS-3 was assessed using an 11-point Numeric Rating Scale (NRS), on this scale 0 indicates no pain and 10 indicates pain as bad as you can imagine. This scale recalls the average pain intensity during the last 3 days. The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your pain on average during the last 3 days (the last 72 hours prior to the visit)".
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 126
units on a scale
  Baseline | 7.7 (1.04) | 7.6 (0.95)
  End of Continuation Period | 3.9 (2.68) | 4.8 (2.43)

4. Secondary Outcome: Change in Recalled Average Pain Intensity at the End of Treatment
Description: The recalled average pain intensity score on the NRS-3 was assessed using an 11-point Numeric Rating Scale (NRS), on this scale 0 indicates no pain and 10 indicates pain as bad as you can imagine. This scale recorded the average pain intensity recalled by the participant during the previous 3 days. The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your pain on average during the last 3 days (the last 72 hours prior to the visit)". A negative sign indicates a decrease in pain from the start of treatment. The higher the absolute values, the greater the change since the start of treatment (baseline visit).
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 126
units on a scale | -3.7 (0.24) | -2.8 (0.24)

5. Secondary Outcome: Average Pain Intensity Over Three Days for Pain Radiating Towards or Into the Leg
Description: Typical dermatomal pain was defined as being pain that radiates beyond the knee towards the foot (sciatica) or pain evoked by stretching of the sciatic nerve.
  The participant was asked to rate their pain intensity over the past 3 days with regards to this particular pain characteristic.
  The recalled average pain intensity over the past 3 days for the pain radiating towards or into the leg was assessed by the participant using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale
  Baseline | 7.5 (1.25) | 7.6 (1.05)
  End of Continuation Period | 3.7 (2.76) | 4.7 (2.52)

6. Secondary Outcome: Change of Average Pain Intensity Over Three Days for Pain Radiating Towards or Into the Leg at the End of Treatment
Description: Typical dermatomal pain was defined as being pain that radiates beyond the knee towards the foot (sciatica) or pain evoked by stretching of the sciatic nerve.
  Therefore, the participant was asked to rate their pain intensity over the past 3 days with regards to this particular pain characteristic.
  The recalled average pain intensity during the last 24 hours was assessed using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
  A negative sign indicates that there was a decrease in the average pain radiating towards or into the leg.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale | -3.9 (0.25) | -2.8 (0.25)

7. Secondary Outcome: Worst Pain Intensity Over the Past 24 Hours
Description: The recalled worst pain intensity during the last 24 hours was assessed using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
  The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your worst pain during the last 24 hours prior to the visit"
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale
  Baseline | 8.1 (1.03) | 8.0 (1.06)
  End of Continuation Period | 4.3 (2.73) | 5.2 (2.50)

8. Secondary Outcome: Change in Worst Pain Intensity Over the Past 24 Hours at the End of Treatment
Description: The recalled worst pain intensity during the last 24 hours was assessed using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
  The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your worst pain during the last 24 hours prior to the visit".
  A negative change indicates that the pain intensity decreased from the start of the trial.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale | -3.7 (0.25) | -2.8 (0.25)

9. Secondary Outcome: painDETECT Final Assessment
Description: The painDETECT was a participant completed questionnaire. The questionnaire consists of 14 questions in four domains. Based on these questions a final assessment score was calculated. The minimum score ranged from zero to a maximum of 38. Participants with a score between 0 and 12 were scored as being "negative" (had no neuropathic pain component). A value between 19 and 38 was rated as being "positive" (neuropathic component present). Values from 13 to 18 were scored as being "unclear". The theoretical range of change in this trial ranged from -38 to 15. A negative change indicated a decrease in their neuropathic component of pain.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 124 | 115
units on a scale
  Baseline | 22.3 (5.25) | 22.5 (4.79)
  End of Continuation Period | 11.9 (7.76) | 14.6 (7.37)

10. Secondary Outcome: Change in painDETECT Final Assessment at the End of Treatment
Description: as for outcome 9
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 124 | 115
units on a scale | -10.8 (0.67) | -7.9 (0.69)

11. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score Assessment
Description: In the Neuropathic Pain Symptom Inventory (NPSI) the participant rated their symptoms of neuropathic pain. Ten pain questions were answered on an 11-point scale; from 0 (symptom not present) to 10 (symptom at its worst imaginable intensity, e.g. worst burning imaginable). The overall NPSI score was calculated by the summation of all ten responses and ranges between 0 and 1. For pain descriptions burning, pressing, paroxysmal (pain like electric shocks or stabbing), evoked (due to touch) and paresthesia (sensation that is not unpleasant) or dysesthesia (unpleasant) sub-scores are reported. The overall values reported for all participants that completed the questionnaire are shown. A symptom was absent if the value is 0, the symptom was present in all participants and all participants rated it at its worst possible intensity if a value is 1.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
units on a scale
  Baseline Overall Score | 0.598 (0.1769) | 0.612 (0.1445)
  End Continuation Period Overall Score | 0.251 (0.2344) | 0.354 (0.2334)
  Baseline Sub-Score Burning Pain | 0.612 (0.2569) | 0.634 (0.2279)
  End Continuation Period Sub-Score Burning Pain | 0.248 (0.2767) | 0.337 (0.2758)
  Baseline Sub-score pressing pain | 0.595 (0.2523) | 0.608 (0.1848)
  End Continuation Period Sub-Score Pressing Pain | 0.276 (0.2650) | 0.375 (0.2645)
  Baseline Sub-Score Paroxysmal Pain | 0.638 (0.2312) | 0.670 (0.1720)
  End Continuation Period Sub-Score Paroxysmal Pain | 0.269 (0.2716) | 0.375 (0.2673)
  Baseline Sub-Score Evoked Pain | 0.555 (0.2536) | 0.548 (0.2300)
  End Continuation Period Sub-Score Evoked Pain | 0.219 (0.2520) | 0.321 (0.2554)
  Baseline Sub-Score Pare/Dysesthesia | 0.621 (0.2292) | 0.642 (0.1809)
  End Continuation Period Sub-Score Pare/Dysesthesia | 0.260 (0.2656) | 0.372 (0.2615)

12. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score Assessment at the End of Treatment
Description: In the Neuropathic Pain Symptom Inventory (NPSI) the participant rated their symptoms of neuropathic pain. Ten pain questions were answered on an 11-point scale, from 0 (symptom not present) to 10 (symptom at its worst imaginable intensity, e.g. worst burning imaginable). The overall NPSI score was calculated by the summation of all ten responses and ranges between 0 and 1. For pain descriptions burning, pressing, paroxysmal (pain like electric shocks or stabbing), evoked (due to touch) and paresthesia (sensation that is not unpleasant) or dysesthesia (unpleasant) sub-scores are reported. The overall values reported for all participants that completed the questionnaire are shown. A symptom was absent if the value is 0, the symptom was present in all participants and all participants rated it at its worst possible intensity if a value is 1. A negative change indicates that the intensity of the symptom has decreased since the start of treatment.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale
  Overall Score | -0.353 (0.0208) | -0.248 (0.0211)
  Sub-Score Burning Pain | -0.375 (0.0249) | -0.278 (0.0252)
  Sub-Score Pressing Pain | -0.331 (0.0235) | -0.226 (0.0238)
  Sub-Score Paroxysmal Pain | -0.385 (0.0246) | -0.283 (0.0250)
  Sub-score Evoked Pain | -0.334 (0.0222) | -0.225 (0.0225)
  Sub-Score Pare/Dysesthesia | -0.363 (0.0229) | -0.252 (0.0231)

13. Secondary Outcome: Short Form Health Survey (SF-12)
Description: The Short Form Health Survey (SF-12) has several brief broad questions on 8 aspects of health (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. The physical and mental summary scores were calculated from the individual responses. A higher score indicates a better participant perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible health state.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
units on a scale
  Baseline Physical Functioning | 33.256 (7.7695) | 33.813 (6.8734)
  End Continuation Period Physical functioning | 41.701 (10.2556) | 39.120 (9.4634)
  Baseline Role-Physical | 33.783 (6.5010) | 33.695 (6.2586)
  End Continuation Period Role-Physical | 41.025 (8.7602) | 38.757 (7.6342)
  Baseline Bodily Pain | 30.430 (7.9923) | 31.117 (8.1434)
  End Continuation Period Bodily Pain | 42.003 (10.1964) | 38.637 (10.3872)
  Baseline General Health | 36.110 (8.3196) | 34.652 (7.0912)
  End Continuation Period General Health | 44.382 (10.3772) | 39.941 (10.1717)
  Baseline Vitality | 46.518 (8.5121) | 45.516 (8.0387)
  End Continuation Period Vitality | 51.202 (9.3262) | 47.724 (10.0303)
  Baseline Social Functioning | 42.290 (10.5832) | 41.734 (9.8674)
  End Continuation Period Social Functioning | 47.494 (10.4657) | 44.475 (10.5281)
  Baseline Role-Emotional | 41.018 (13.0098) | 37.046 (13.2164)
  End Continuation Period Role-Emotional | 44.727 (12.1390) | 41.219 (12.7890)
  Baseline Mental Health | 44.967 (9.2036) | 42.394 (9.1589)
  End Continuation Period Mental health | 49.828 (10.3896) | 46.451 (10.3372)
  Baseline Physical Component summary | 30.319 (7.2739) | 31.684 (6.8313)
  End Continuation Period Physical component summary | 40.493 (9.3352) | 37.765 (8.8375)
  Baseline Mental Component Summary | 48.736 (11.5697) | 45.216 (11.7462)
  End Continuation Period Mental Component Summary | 51.117 (11.0365) | 47.595 (11.4544)

14. Secondary Outcome: Changes in the Short Form Health Survey (SF-12) at the End of Treatment
Description: The Short Form Health Survey (SF-12) has several brief broad questions on 8 aspects of health (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. The physical and mental summary scores were calculated from the individual responses. A higher score indicates a better participant perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible health state.
  The change in the SF-12 score shows an improvement in health from baseline if the values are positive. The higher the value the greater the improvement since starting the trial.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS), Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale
  Physical Functioning | 8.358 (0.8262) | 5.073 (0.8361)
  Role-Physical | 7.260 (0.7115) | 4.668 (0.7224)
  Bodily Pain | 10.990 (0.9462) | 7.458 (0.9570)
  General Health | 8.447 (0.8702) | 4.309 (0.8818)
  Vitality | 4.943 (0.8062) | 1.468 (0.8179)
  Social Functioning | 5.246 (0.8870) | 2.286 (0.8997)
  Role-Emotional | 4.764 (0.9472) | 2.587 (0.9807)
  Mental Health | 5.158 (0.8386) | 2.973 (0.8575)
  Physical Component Summary | 9.735 (0.7948) | 6.202 (0.8058)
  Mental Component Summary | 3.077 (0.8457) | 1.146 (0.8679)

15. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome
Description: The participant scored the EuroQol-5 questionnaire. The EuroQol-5 questionnaire uses a health state classification with 5 dimensions. Each dimension was assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1 (with 1 indicating "full health" and 0 representing "dead"). The higher the values (the closer the value is to 1) the better the health status in a treatment group.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
units on a scale
  Baseline | 0.3186 (0.29464) | 0.3392 (0.31134)
  End of Continuation Period | 0.6686 (0.31683) | 0.5745 (0.31378)

16. Secondary Outcome: Change in EuroQol-5 (EQ-5D) Health Status Index Outcome at the End of Treatment
Description: as for outcome 15
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
units on a scale | 0.3395 (0.02785) | 0.2398 (0.02811)

17. Secondary Outcome: Hospital Anxiety and Depression Scale: Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate anxiety. A score of 11 or above is considered to be a case of anxiety.
  A decrease in values over the trial period indicate that there has been an improvement.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 124
units on a scale
  Baseline | 7.3 (4.06) | 8.2 (4.28)
  End of Continuation Period | 5.3 (4.40) | 6.7 (4.58)

18. Secondary Outcome: Change in Hospital Anxiety and Depression Scale at the End of Treatment: Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate anxiety. A score of 11 or above is considered to be a case of anxiety.
  A negative sign indicates that there has been a decrease in anxiety since the start of treatment.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 124
units on a scale | -2.1 (0.34) | -1.1 (0.35)

19. Secondary Outcome: Hospital Anxiety and Depression Scale: Depression
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe depression. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate depression. A score of 11 or above is considered to be a case of depression. A decrease in values over time indicates that there has been an improvement.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last observation carried forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
units on a scale
  Baseline | 7.4 (4.08) | 8.0 (4.08)
  End of Continuation Period | 5.1 (4.17) | 6.5 (4.86)

20. Secondary Outcome: Change in Hospital Anxiety and Depression Scale at the End of Treatment: Depression
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe depression. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate depression. A score of 11 or above is considered to be a case of depression. A decrease in values over time indicates that there has been an improvement. A negative change value indicates a decrease in the depression score since the start of treatment.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last observation carried forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 124 | 114
units on a scale | -2.4 (0.34) | -1.1 (0.36)

21. Secondary Outcome: Patient Global Impression of Change at the End of Treatment
Description: In the Patient Global Impression of Change (PGIC) the participant indicated the perceived change over the treatment period. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 129 | 125
participants
  Very Much Improved | 27 | 18
  Much Improved | 43 | 19
  Minimally Improved | 32 | 46
  No Change | 21 | 29
  Minimally Worse | 3 | 6
  Much Worse | 2 | 4
  Very Much Worse | 1 | 3

22. Secondary Outcome: Clinician Global Impression of Change at the End of Treatment
Description: In the Clinician Global Impression of Change (CGIC) the clinician indicated the perceived change over the treatment period. The clinician was requested to choose one of seven categories for each participant. The Clinician rated the participants change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 128 | 123
participants
  Very Much Improved | 32 | 18
  Much Improved | 44 | 25
  Minimally Improved | 22 | 37
  No Change | 21 | 26
  Minimally Worse | 6 | 7
  Much Worse | 3 | 9
  Very Much Worse | 0 | 1

23. Secondary Outcome: Sleep Evaluation at the End of Treatment: Change in the Overall Quality of Sleep
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the overall quality of sleep.
  The participant rated this categorically as being one of the following: excellent, good, fair or poor.
  The improvement, no change or worsening is reported based on the replies scored by the participants given at their End of Continuation Visit.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 126
participants
  Improvement | 62 | 43
  No Change | 46 | 56
  Worsening | 16 | 15
  Missing | 6 | 12

24. Secondary Outcome: Sleep Evaluation: Number of Awakenings
Description: The participants were requested to answer the following question:
  How many times did you wake up during the night? The values were calculated from the data that participants self-reported for the night prior to their Randomization Visit (Baseline) and for the night prior to the End of the Continuation Visit (12 weeks after randomization).
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
number of awakenings
  Baseline | 3.0 (2.80) | 2.6 (1.67)
  End of Continuation Period | 2.0 (1.66) | 2.2 (1.65)

25. Secondary Outcome: Sleep Evaluation at the End of Treatment: Change in the Number of Awakenings
Description: The participants were requested to answer the question: How many times did you wake up during the night? The values were calculated from the data that participants self-reported. The change from baseline in the number of times of waking up during the night in a treatment group is reported. A negative symbol indicates that there was a reduction in the number of awakenings.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF). Number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 124 | 114
number of awakenings | -0.8 (0.15) | -0.5 (0.16)

26. Secondary Outcome: Sleep Evaluation: Number of Hours Slept
Description: The participants were requested to answer the following question:
  How long did you sleep last night [hours]? The values were calculated from the data that participants self-reported for the night prior to their Randomization Visit (Baseline) and for the night prior to the End of the Continuation Visit (12 weeks after randomization).
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 125
hours
  Baseline | 5.781 (1.5908) | 5.675 (1.7118)
  End of Continuation Period | 6.207 (1.8007) | 6.218 (1.8426)

27. Secondary Outcome: Sleep Evaluation at the End of Treatment: Change in the Number of Hours Slept
Description: The sleep evaluation questionnaire was completed by the participant. The answer was in response to the question: Sleep evaluation: How long did you sleep last night [hours]? The value reported is the change in the number of hours of sleep from baseline. The positive value indicates that there was an increase in the number of hours of sleep in a treatment group.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS). Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 126
hours | 0.460 (0.1714) | 0.412 (0.1763)

28. Secondary Outcome: Sleep Evaluation: Latency (Time Taken to Fall Asleep)
Description: The sleep evaluation questionnaire was completed by the participant. The participant was asked: How long after bedtime/lights out did you fall asleep last night [hours]? The values are for the night prior to the Randomization Visit (Baseline) and for the night prior to the Final Evaluation Visit (12 weeks after randomization). The higher the value the longer it took to fall asleep.
Time Frame: Baseline (Randomization Visit); End of Continuation Period (Week 12)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Oxycodone/Naloxone Prolonged Release: All participants started with 10 mg/5 mg oxycodone/naloxone prolonged release (twice daily). The dose of oxycodone/naloxone prolonged release could be adjusted in increments of 10mg/5 mg oxycodone/naloxone to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 50 mg/20 mg oxycodone/naloxone twice daily (100 mg/40 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 126
hours
  Baseline | 1.047 (1.1746) | 1.203 (1.3029)
  End of Continuation Period | 0.803 (1.1154) | 0.865 (1.0301)

29. Secondary Outcome: Sleep Evaluation at the End of Treatment: Change in Latency (Change in the Time Taken to Fall Asleep)
Description: The sleep evaluation questionnaire was completed by the participant. The participant was asked: How long after bedtime/lights out did you fall asleep last night [hours]? The values are for the night prior to the visits. The negative change from baseline indicates that the time to falling asleep decreased from baseline in a treatment group.
Time Frame: Baseline (Randomization Visit); End of Continuation Visit (Week 12)
Population: Full Analysis Set (FAS). Last Observation carried Forward (LOCF). Number of participants taken into account for the analyses.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 124 | 114
hours | -0.300 (0.1000) | -0.177 (0.1025)

30. Secondary Outcome: Comparison of the Number of Participants Affected by Gastrointestinal Treatment Emergent Adverse Events (TEAEs) Typical for Opioids
Description: In this outcome measure the number of participants affected by early gastrointestinal-related treatment emergent adverse events (TEAEs). As the trial population was opioid-naïve this was considered of interest.
  The composition score from participant who reported:
  Mild, moderate to severe nausea and/or Mild, moderate to severe vomiting and/or Mild, moderate to severe constipation was evaluated.
Time Frame: Baseline (Randomization Visit) to End of Titration Period (End of Week 3)
Population: Safety Set (SAF).
Measure: Number; unit: participants
Groups:
- Oxycodone/Naloxone Prolonged Release: All participants started with 10 mg/5 mg oxycodone/naloxone prolonged release (twice daily). The dose of oxycodone/naloxone could be adjusted in increments of 10 mg/5 mg oxycodone/naloxone to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 50 mg/20 mg oxycodone/naloxone twice daily (100 mg/40 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 128
participants | 42 | 59

31. Secondary Outcome: Composite Event Based Comparison of Gastrointestinal Treatment Emergent Adverse Events (TEAEs) Typical for Opioids
Description: In this outcome measure the early gastrointestinal-related treatment emergent events (TEAEs) were evaluated. As the trial population was opioid-naïve this was considered of interest.
  The composition score of reported events of Mild, moderate to severe nausea and/or Mild, moderate to severe vomiting and/or Mild, moderate to severe constipation was evaluated.
Time Frame: Baseline (Randomization Visit); End of Week 3 (End of Titration Period)
Population: Safety Set (SAF).
Measure: Number; unit: number of events
Arm/Group | Tapentadol Prolonged Release | Oxycodone/Naloxone Prolonged Release
Number analyzed (Participants) | 130 | 128
number of events | 56 | 81

ADVERSE EVENTS:
Time Frame: Adverse events occurring after first administration of study drug were listed (Treatment emergent adverse events - TEAEs) and within 3 days after the last intake were considered as TEAEs. Pre-treatment adverse events that worsened were considered TEAEs.
Groups:
- Tapentadol Prolonged Release (PR): All participants started with 50 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted in increments of 50 mg to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
- Oxycodone/Naloxone Prolonged Release (PR): All participants started with 10 mg/5 mg oxycodone/naloxone prolonged release (twice daily). The dose of oxycodone/naloxone prolonged release could be adjusted in increments of 10 mg/5 mg oxycodone/naloxone to a level that provided adequate analgesia. The next titration step was after a minimum of 3 days on a dose. Participants were permitted a maximum dose of 50 mg/20 mg oxycodone/naloxone twice daily a day (100 mg/40 mg total daily dose). After titration participants remained on the stable dose for 9 weeks.
- Tapentadol (PR) After Oxycodone/Naloxone (PR) Treatment: Participants in the oxycodone/naloxone PR treatment arm that did not reach the minimum target of titration or experiencing intolerable side effects at the end of the Titration Period could be switched to the Pick-up Arm. They could also enter the Pick-up Arm at any time during the Titration Period or Continuation Period, via an unscheduled visit, due to lack of tolerability or lack of efficacy under treatment with oxycodone/naloxone PR. Participants were directly switched from oxycodone/naloxone PR to tapentadol PR using an equianalgesic ratio of 1:5 (oxycodone : tapentadol), together with a down-titration step under tapentadol PR (except for participants on oxycodone/naloxone PR 10 mg/5 mg twice daily).
Arm/Group | Tapentadol Prolonged Release (PR) | Oxycodone/Naloxone Prolonged Release (PR) | Tapentadol (PR) After Oxycodone/Naloxone (PR) Treatment
Serious Adverse Events (participants affected / at risk) | 3/130 | 2/128 | 0/50
Other Adverse Events (participants affected / at risk) | 97/130 | 105/128 | 29/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapentadol Prolonged Release (PR) (N=130) | Oxycodone/Naloxone Prolonged Release (PR) (N=128) | Tapentadol (PR) After Oxycodone/Naloxone (PR) Treatment (N=50)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapentadol Prolonged Release (PR) (N=130) | Oxycodone/Naloxone Prolonged Release (PR) (N=128) | Tapentadol (PR) After Oxycodone/Naloxone (PR) Treatment (N=50)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 5 (6) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (20) | 33 (34) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 7 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (31) | 23 (23) | 5 (7)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (11) | 21 (24) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 39 (42) | 31 (32) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (3) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (5) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Biopsy chest wall (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 24 (26) | 22 (22) | 6 (6)
Headache (Nervous system disorders) | 10 (10) | 5 (5) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 5 (6) | 1 (1)
Neuromuscular blockade (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Vertigo cns origin (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (2) | 2 (2) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8) | 13 (13) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 11 (12) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 7 (7) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.